CLINICAL TRIAL: NCT06605963
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study Evaluating the Safety and Efficacy of PPV-06 Active Immunotherapy in Patients With Inflammatory Knee Osteoarthritis (KOA)
Brief Title: PPV-06 Vaccine in Inflammatory Knee Osteoarthritis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peptinov SAS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PPV-06-KOA-201; 2024-514388-24 (EudraCT Number)
Record Dates: First submitted 2024-05-31; First posted 2024-09-20 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Osteoarthritis, Knee
Keywords: Inflammatory osteoarthritis; Immunotherapy; Interleukine-6
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Randomized, Parallel Group, Double-Blind, Placebo-Controlled, Multicenter Study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PPV-06 (Experimental): PPV-06 10 μg + Montanide™ ISA 51 VG in subcutaneous administration
  Interventions: Drug: PPV-06
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PPV-06 — 6 subcutaneous injections at Day 1, Week 4, Week 24, Week 44, Week 64, Week 84
  Arms: PPV-06
Drug: Placebo — 6 subcutaneous injections at Day 1, Week 4, Week 24, Week 44, Week 64, Week 84
  Arms: Placebo

SUMMARY:
PPV-06 targets interleukin-6, a key molecule implicated in many inflammatory diseases such osteoarthritis. PPV-06 is used to induce the production of antibodies directed against IL-6. The antibodies produced will neutralize the interleukine-6 involved in the body's inflammatory process.

The goal of this clinical trial is to test the safety and efficacy of PPV-06 in participants with Knee Osteoarthritis. The main questions are to evaluate if PPV-06 can reduce pain and improve functioning in participants with knee osteoarthritis, and to evaluate if ¨PPV-06 is safe when administered to participants.

Participants will be administered with 6 subcutaneous injections of either PPV-06 or placebo, over a two-year period.

DETAILED DESCRIPTION:
This study assesses the safety and efficacy of PPV-06 active immunotherapy versus placebo in patients who have inflammatory osteoarthritis of the knee.

PPV-06 active immunotherapy will be assessed at a dose level of 10 µg. In total, 204 patients will be randomized to receive either IMP or placebo in a ratio 1:1.

Patients will each receive 6 injections of IMP or a placebo during the Double-blind Treatment Period of 104 weeks. For each SC injection, patients will receive the same IMP or Placebo that was administered at the first injection, in a double-blind manner.

The study comprises a total of 13 scheduled on site visits and 5 scheduled phone calls, which are considered appropriate to collect trial data, monitor patients' safety, and support patients' compliance to meet trial objectives.

The overall study duration by patient will be approximately 108 weeks (up to 4 weeks for screening visit and 104 weeks of study treatment). The study comprises:

* Screening period - V1 (up to - 28 days);
* Treatment induction immune response period - V2 (D1), V3 (W4), V4;
* Maintenance immune response period - V5 (W24), V6, V7 (W44), V8, V9 (W64), V10, V11 (W84), V12 ;
* Phone calls between each scheduled visits as per protocol (PC1, PC2, PC3, PC4, PC5);
* End of Study visit or Early Termination visit - V13 (W104).

Efficacy evaluations, including pain and physical function assessments, MSK examinations, MRI with contrast, clinical laboratory tests and health related quality of life (such as WOMAC, NRS, PGA, SF-36, EQ-5D-5L, PGIC, PSQI, PSFS, WPAI questionnaires by e-PRO and e-Diary) will be performed.

Safety evaluations, including physical examinations, vital signs, ECGs, X-Ray, Ultrasound (US), MRI with contrast, and clinical laboratory tests will be performed.

Concomitant medication usage will be recorded from the time of screening until the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant has given written informed consent to participate.
* Male or female, aged at least 40 years old.
* BMI between 22 to 35kg/m² at Screening visit.
* Diagnosis of osteoarthritis of the index knee based on American College of Rheumatology (ACR) criteria and functional capacity class of I-III, with a Kellgren-Lawrence grade [KLG] 2 or 3.
* OARSI medial Joint Space Narrowing (mJSN) Grade 1 or 2 of the index knee joint, confirmed by a semi-flexed or fixed flexion weight-bearing X-Ray performed at Screening visit, and assessed by Central Reader.
* Evidence during the Screening visit of synovitis in the index knee based on ultrasound as described in the Ultrasound Doppler manual.
* Evidence of moderate to severe Synovitis on 11-point synovitis (based on Guermazi et al. score), as assessed by Rapid OA MRI Eligibility Score (ROAMES(1)), per-formed during the Screening visit and assessed by Central Reader.
* Insufficient pain relief with standard of care (i.e. non-pharmacological treat-ments, systemic non-steroidal anti-inflammatory drugs (NSAIDs) and/or other analgesics) for symptomatic OA in the index knee within 6 months prior to the Screening vis-it.
* Pain at index knee for the majority of days (>50%) during the preceding month prior to the Screening Visit.
* At Screening Visit 1a, participant reports that their typical OA knee pain in one or both knees when not using medication is ≥ 4 out of 10.
* WOMAC pain subscale score (5 items) in the range [≥4 and ≤8], using the 11-point (0-10) NRS for the index knee at Screening and Baseline visits.
* Participant is willing to discontinue all pain medications for OA except rescue medication (pa-racetamol), to adhere to the restricted use of concomitant treatments and not use prohibited pain medications throughout the clinical trial.

Exclusion Criteria:

* Participant had an administration of NSAID (topical, tablets) or Cox-2 Inhibitors within 2 weeks prior to the Baseline visit.
* Injection of either corticosteroid or intra-articular (IA) Visco-supplementation (i.e., hyaluronic acid) into the index knee within 1 month of Screening.
* Injection of platelet-rich plasma (PRP) into the index knee within 6 months of Screening.
* Application of topical capsaicin on the index knee within 1 month of Screening.
* Past joint replacement surgery of the index knee.
* History of significant trauma or surgery (e.g., open or arthroscopic) to the in-dex knee within 12 months of Screening.
* Scheduled surgery except dental surgery during the clinical trial period.
* Any known active infection, including suspicion of intra-articular infection, ul-cer or open wound anywhere on the index knee.
* Periarticular pain from any cause other than osteoarthritis, including referred pain, bursitis, tendinitis, soft tissue tenderness, or subacute/acute pain from injury in the index knee.
* Known presence of pre-existing MRI-based findings warranting exclusion in accordance with the ROAMES criteria, such as rapidly progressing osteoarthritis (RPOA) Type I or Type II, osteonecrosis, subchondral insufficiency fracture, atrophic oste-oarthritis, severe bone on bone osteoarthritis, or knee pain attributable to disease other than osteoarthritis, or as assessed by X-Ray, based on Central imaging Reading at Screening Visit and before the Baseline Visit.
* Significant malalignment of anatomical axis (medial angle formed by the femur and tibia) of the index knee (varus >10°, valgus >10°) by X-Ray as assessed by Central Readers at Screening Visit.
* Other conditions that could affect trial endpoint assessments of the index knee, including, but not limited to, rheumatoid arthritis, psoriatic arthritis, ankylosing spondyli-tis, gout or pseudogout, inflammatory bowel disease related arthropathy, peripheral neuropathy, lupus erythematosus, significant skin conditions such as abscesses, acromegaly, metabolic joint diseases and fibromyalgia.
* Neuropathic pain as assessed by PainDETECT questionnaire with a score of at least 18 at Screening Visit.
* Systemic (except inhaled) immunosuppressant agent within 6 months prior to trial medication administration.
* Current clinically significant disease(s) or condition(s) (including clinically significant cardiovascular disease and/or significant pain in other areas) that may affect efficacy or safety assessments, or any other reason which, in the investigator's opinion, may preclude the patient's participation in the full duration of the trial.
* Major bleeding disorder encompassing, but not limited to coagulopathy and any current antithrombotic and anticoagulant events.
* History of severe allergic or anaphylactic reactions.
* Known infection of human immunodeficiency virus (HIV), or known current acute or chronic hepatitis B or C infection.
* Unstable or poorly controlled blood pressure which, in the opinion of the inves-tigator, would put the patient at risk of severe adverse blood pressure increases upon IMP administration.
* History of malignancy within 5 years prior to the Screening visit, with the ex-ception of basal cell carcinoma.
* History of either active TB or latent TB with inadequate course of anti-tuberculous prophylaxis.
* Contraindications to an MRI (including the gadolinium contrast with a Glo-merular Filtration Rate (GFR) below 60 mL/min) of the index knee or has a pacemaker or any other implanted electronic devices. Claustrophobic patient with impossibility to under-go an MRI.
* Evidence or history of severe psychiatric illness/disorder during 3 years prior to the Screening Visit that, in the investigator's opinion, may affect safety or efficacy assess-ments or may compromise the patient's safety during trial participation.
* Known or suspected of not being able to comply with the requirements of the trial protocol or the instructions of the trial site staff.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of PPV-06 on pain in participants with knee Osteoarthritis | From Baseline to Week 54
  Absolute change from baseline to Week 54 of the pain subscale score of the Western Ontario and McMaster University scale (WOMAC)
To evaluate the efficacy of PPV-06 on physical functioning in participants with knee Osteoarthritis | From Baseline to Week 54
  Absolute change from baseline to Week 54 of the Western Ontario and McMaster University (WOMAC) physical function subscale score

SECONDARY OUTCOMES:
To evaluate the efficacy of PPV-06 on key structural features of knee Osteoarthritis | From Baseline to Week 104
  Absolute change from baseline in cartilage thickness (ThC) in the medial femorotibial compartment (MFTC)
Cartilage thickness | From Baseline to Week 104
  Absolute change from baseline in cartilage thickness (ThC) assessed by MRI at 1 and 2 years (W54 and W104) using quantitative image analysis method
Safety and Tolerability of PPV-06 | From Baseline to Week 104
  Incidence of Adverse Events of Special Interest (AESI).
To evaluate the efficacy of PPV-06 on key inflammation features of knee Osteoarthritis | From Baseline to Week 54
  Absolute Change from baseline to Week 54 of Synovitis based on Rapid OsteoArthritis MRI Eligibility Score (ROAMES) 11-point synovitis score
Western Ontario and McMaster University total score | From baseline to Week 54
  Absolute Change of the Western Ontario and McMaster University (WOMAC) total score

OTHER OUTCOMES:
Immune response and development of antibodies to treatment with PPV-06 | From Baseline to Week 104
  Change from baseline in inflammatory markers in serum (Il-6, hsCRP, CRPM)

CONTACTS AND LOCATIONS:
Locations (1):
- CIC Cochin, Paris, France

IPD SHARING:
Plan to Share IPD: No